CLINICAL TRIAL: NCT06312917
Title: Effects of Physical Activity Based on the Transtheoretical Model on Patients With Endometrial Cancer Undergoing Fertility-sparing Treatment: a Randomized Controlled Trial
Brief Title: Effect of Physical Activity Intervention on Overweight and Obese Patients With Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Li, associate professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023PHB183
Record Dates: First submitted 2024-02-25; First posted 2024-03-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Endometrium Cancer; Physical Activity; Weight Management
MeSH Terms: conditions — Endometrial Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity group (Experimental): Exercise intervention According to the guidelines of the American Sports Medicine Association (ACSM) and the National Fitness guidelines of the General Administration of Sport of China
  Interventions: Behavioral: Physical activity
- control group (No Intervention): Maintain the current state of physical activity, do not do physical activity intervention.

INTERVENTIONS:
Behavioral: Physical activity — Exercise intervention According to the guidelines of the American Sports Medicine Association (ACSM) and the National Fitness guidelines of the General Administration of Sport of China, the FITT-VP principle of ACSM is adopted. The patients were given the intervention guidance of aerobic exercise, resistance training and flexibility training. During the training, the patients filled in the weekly training records, including the feeling after each training, physical dimension and other relevant information, and the nurses gave personalized exercise guidance according to the patients' conditions.The diet is to maintain a balanced diet.
  Arms: Physical activity group

SUMMARY:
This study evaluated the clinical outcome of exercise management on patients with endometrial cancer treated with fertility preservation, including the effect of complete response rate, complete response time, recurrence rate, recurrence time, etc., and physical composition, to evaluate the effectiveness of physical activity on weight management.

ELIGIBILITY:
Inclusion Criteria:

* Participants were patients who met the following predefined eligibility criteria: Ages 20-40; Overweight or obese; The pathological diagnosis was EC (endometrioid, grade I, no myometrium invasion or metastasis). Not pregnant; Be willing to comply with test requirements after being fully informed of all risks and inconveniences associated with the test.

Exclusion Criteria:

* Recurrent or metastatic disease; Currently participating in regular exercise at least 2 days per week; Pregnant at the start of the study; Or unwilling to comply with research requirements. Patients also completed the Physical Activity Readiness Questionnaire (PAR-Q) through a telephone interview. Patients with one or more potential exercise-related safety risks were excluded.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Body weight | Enrollment，four months after the intervention
  Body weight measured naked or wearing work clothes of known weight, an electronic weight scale is used to measure
BMI | Enrollment，four months after the intervention
  Body mass index is a standard commonly used in the world to measure the degree of body fat and whether it is healthy.
  The formula is BMI= weight ÷ height*height
physical activity level | Enrollment，four months after the intervention
  Physical activity energy was calculated using the formula of the International Physical Activity Questionnaire. Calculation Manual: Physical activity amount (MEt-minutes /week)= physical activity intensity MET value × physical activity time (minutes)/ day × activity days.

SECONDARY OUTCOMES:
serum total cholesterol | Enrollment，four months after the intervention
  Total cholesterol is the sum of all lipoproteins in the blood.The measurement was made by drawing venous blood. Suitable level for adults: 2.83~5.20mmol/L(110~200mg/dl)
Waist Hip Ratio | Enrollment，four months after the intervention
  It is an indicator of the distribution of human body fat. It is the ratio of the waist and abdomen circumference marked by the umbilicus to the hip circumference marked by the anterior superior spine of the iliac (cm).
triglyceride | Enrollment，four months after the intervention
  Serum triglyceride determination is a routine item in lipid analysis. The measurement was made by drawing venous blood. Normal reference value of serum triglyceride: 0.45 ~ 1.69mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided